CLINICAL TRIAL: NCT06265077
Title: Efficacy and Safety of Loratadine and Famotidine Combination on Preventing Filgrastim-Induced Bone Pain in Breast Cancer Patients
Brief Title: Novel Preventive Approach Against Filgrastim-Induced Bone Pain in Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Noha Mansour (Other)
Responsible Party: Sponsor-Investigator, Noha Mansour, Lecturer of Clinical Pharmacy-Clinical Pharmacy and Pharmacy Practice Department, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2023-199
Record Dates: First submitted 2024-02-10; First posted 2024-02-20 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Filgrastim Adverse Reaction
MeSH Terms: conditions — Breast Neoplasms | interventions — Famotidine; Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): (intervention group) patients who will receive filgrastim plus oral famotidine 20 mg once daily and loratadine 10 mg once daily for the full filgrastim treatment period.
  Interventions: Drug: famotidine and loratadine
- Control (Placebo Comparator): (control group) patients who will receive placebo plus filgrastim.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Control
Drug: famotidine and loratadine — famotidine 20 mg once daily and loratadine 10 mg once daily
  Arms: Intervention

SUMMARY:
No randomized controlled trial evaluated the safety and efficacy of double blockade on G-CSF induced bone pain. Therefore, this study aims to evaluate the efficacy and safety of double blockade on the incidence and severity of G-CSF induced bone pain.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients were 18 years or older.
2. Confirmed diagnosis of breast cancer.
3. Patients completed adriamycin and cyclophosphamide (AC) regimen and are planned to receive four cycles or more of paclitaxel chemotherapy with G-CSF support starting in cycle 1 and continuing throughout each of the four paclitaxel cycles.
4. Eastern Cooperative Oncology Group (ECOG) performance status from 0 to 2.

Exclusion Criteria:

1. Patients with signs and symptoms of grade 2 or 3 bone pain at baseline.
2. Patients receiving famotidine in the previous 72 hours.
3. Patient receiving any antihistaminic in the previous 72 hours.
4. Hypersensitivity to famotidine or loratadine.
5. Patient receiving opioid or adjuvant analgesic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
The incidence of grade 2 or 3 bone pain in cycle 1 according to Common Terminology Criteria for Adverse Events | two weeks
  Difference between the two arms regarding the incidence of grade 2 or 3 bone pain in cycle 1 according to Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Province, Egypt

IPD SHARING:
Plan to Share IPD: Undecided